CLINICAL TRIAL: NCT02606201
Title: Peri-sphincter Injection of Autologous Myofibres to Treat of Urinary Incontinence by Sphincter Deficiency
Acronym: IPSMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P130927
Record Dates: First submitted 2015-10-20; First posted 2015-11-17 (Estimated); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Urinary Incontinence by Intrinsic Sphincter Deficiency
Keywords: stress urinary incontinence; intrinsic sphincter deficiency; myofiber; autologous; skeletal muscle precursor cells; autologous serum
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IPSMA (Experimental): Injection Peri Sphincter Myofibers Autologous
  Interventions: Other: Peri sphincter injection Autologous myofibers

INTERVENTIONS:
Other: Peri sphincter injection Autologous myofibers — The first step of the procedure consists to harvest a muscle fragment from the lower part of the rectus abdominis muscle of the abdomen approached by a short incision. Injectable myofiber cores will be prepared by hydrodissection of the muscle biopsy.
  All myofibers cores will be suspended in autologous serum prepared by centrifugation before the incision.
  During the second step of the procedure, the myofibers will be injected percutaneously into the peri-sphincter region under endoscopic and radiographic control.

SUMMARY:
Stress urinary incontinence related to intrinsic sphincter deficiency (ISD) is a severe form of incontinence that may have a major impact on the quality of life. The main treatment is surgical and consists in the implantation of medical devices such as the artificial urinary sphincter, adjustable continence therapy, compressive sling, or injection of bulking agent.

The investigator has developed a new therapeutic strategy for ISD that consist to implant myofibers with their attached satellite cells (the main source of muscle progenitor cells) at the vicinity of the striated urethral sphincter. The principle of this method relies on the in vivo activation of satellite cells leading to the formation of regenerated myofibers (myotubes) generating a distinct and tonic muscular activity . The proof of concept was investigated in a Phase I clinical trial: Investigator found that the periurethral implantation of myofiber strips around the urethra generated an electromyographic activity improving urethral closure pressure in women with severe urinary incontinence associated to ISD. In this previous study, the technique of myofiber implantation was invasive, as it required a surgical approach and dissection of the urethra to place the myofiber. For the clinical trial IPSMA, the investigator sought to optimize the myofiber transplantation process using a method injection of myofibers core obtained by hydro-dissection. The injection technique is performed percutaneously under fluoroscopic and endoscopic control and does not require a surgical approach of the urethra.

This clinical trial is prospective, open-label, non-randomized, uncontrolled, single-center for the first stage and multicenter for the second stage, of 13 months for each patient aims to assess the efficacy and safety of IPSMA in the treatment of urinary incontinence in women with ISD.

DETAILED DESCRIPTION:
The investigator chose an assessment method in 2 stages according to the Simon plane . A total of 38 patients are needed. Assuming a ratio of 10% of lost patients or for which the primary endpoint was not evaluable, 4 additional patients will be included totaling 42 patients will be included.

This trial is single-center for the first stage and multicenter for the second stage.

11 patients will be included in the first stage and 31 patients in the second stage.

ELIGIBILITY:
Inclusion Criteria:

* Female.
* Age> or = 18 years.
* Patients with stress urinary incontinence by ISD for at least 6 months Failure of Pelvic ﬂoor muscle training (at least 20 sessions).
* Fixed urethra : a negative Ulmsten test / Qtip test <30 °
* 24h Pad test >50 g
* Urodynamic criteria: LPP (leak points pressure) <100 cm H20 and MUCP <50 cm H2O replaced by Urodynamic criteria: MUCP <50 cm H2O (amendment n°3)
* Collection of informed written consent

Exclusion Criteria:

* Not affiliated to a social security scheme
* Trouble hemostasis known
* Untreated urinary tract infection
* Muscle disease genetically determined or acquired
* Patients with urinary incontinence by vesica-urethral hypermobility
* Incomplete bladder emptying: post void residual> 20% of the volume voided during urination> 150cc
* Maximum urinary flow rate <12 ml / sec replaced by maximum urinary flow rate <12 ml / sec for volume urinated during urination > 150cc (amendment n°3)
* overactive bladder
* Bladder capacity (B3) <200 cc (deleted in amendment n°3)
* Urethral stricture
* Anticoagulant therapy that cannot be replaced by a low molecular weight heparin
* Pregnant or intend to become pregnant during the study period or breastfeeding informed by the patient during the consultation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
Step 1: Tolerance | One year after treatment
  - Tolerance: Serious adverse events grade 3 or more related to the procedure according to Data Safety and Monitoring Board (DSMB)
Step 1 and 2: Rate of patients responder at M12 after surgery | One year after treatment
  Efficiency: Response is defined by an improvement in 24h pad weight as greater than 50% reduction from baseline and improvement in the number of incontinence episodes per day as greater than 50% reduction from baseline

SECONDARY OUTCOMES:
Occurrence of serious and non-serious adverse events | One year after treatment
Proportion of patients cured at M12. patients are considered as cured if: - The absence of pad use, a 24h pad test <2g AND - The absence of urinary leakage reported in the voiding diary (3 consecutive days). | One year after treatment
Improvement of quality of life | One year after treatment
Response times | One year after treatment
Urodynamic evaluation | One year after treatment
  Leak Point Pressure (LPP), maximal urethral closure pressure (MUCP), area under the curve (profilometry), electromyogram (EMG) gives urodynamic evaluation
Number of re-intervention required (conventional treatment after 6 months) to treat persistent urinary incontinence after IPSMA | 6 months after treatment
Patients with a reduction in the 24h pad test <50% at one year will be considered failure. | One year after treatment
Direct global cost of IPSMA surgery | One year after treatment
Healing times | One year after treatment
  Defined by :
  * The absence of pad use, a 24h pad test <2g AND
  * The absence of urinary leakage reported in the voiding diary (3 consecutive days).

CONTACTS AND LOCATIONS:
Overall Officials: René YIOU, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWNED BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION

REFERENCES:
- [Result] Yiou R, Hogrel JY, Loche CM, Authier FJ, Lecorvoisier P, Jouany P, Roudot-Thoraval F, Lefaucheur JP. Periurethral skeletal myofibre implantation in patients with urinary incontinence and intrinsic sphincter deficiency: a phase I clinical trial. BJU Int. 2013 Jun;111(7):1105-16. doi: 10.1111/j.1464-410X.2012.11682.x. Epub 2013 Mar 7. PMID 23470219